CLINICAL TRIAL: NCT05615649
Title: Expanded Indications in the Pediatric BONEBRIDGE Population
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G220197
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Conductive; Hearing Loss, Mixed
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Study procedure (Experimental): This single-arm, repeated-measures study includes study visits at baseline, surgery, device activation, and at 1, 3, 6, and 12 months post-activation.
  Interventions: Device: MED-EL BONEBRIDGE Bone Conduction Implant

INTERVENTIONS:
Device: MED-EL BONEBRIDGE Bone Conduction Implant — Subjects will be implanted with the MED-EL BONEBRIDGE Bone Conduction Implant System. Subjects will be fit with the appropriate external audio sound processor.
  Other Names: BCI 602

SUMMARY:
This study will assess safety and efficacy of the MED-EL BONEBRIDGE Bone Conduction Implant in children under 12 years old with conductive or mixed hearing loss.

DETAILED DESCRIPTION:
This prospective multicenter IDE study will include 36 children implanted with the MED-EL BONEBRIDGE system at six academic medical centers across the US.

ELIGIBILITY:
Inclusion Criteria:

* Under 12 years of age
* Unaided bone-conduction thresholds at 0.5, 1, 2, and 4 kHz better than or equal to 45 dB HL in the ear to be implanted
* Sufficient air-bone gap (ABG) at in the ear to be implanted
* HRCT scan that confirms sufficient bone quantity and quality to recess and fix the BCI in the ear to be implanted
* Developmental, cognitive, and language skills needed to provide an unaided speech recognition threshold (SRT) in quiet with English spondees
* Prior experience with acoustic or bone conduction hearing aids, unless candidate is unable to wear amplification for medical reasons
* Parental commitment to comply with all study procedures

Exclusion Criteria:

* Children under 3 years (36 months) of age
* Chronic or non-revisable vestibular or balance disorders
* Abnormally progressive hearing loss
* Prior use of a hearing implant in the ear to be implanted
* Current/ongoing use of a hearing implant in the contralateral/non-implant ear
* Evidence that hearing loss is retrocochlear in origin
* Medical condition that contraindicates implant surgery or anesthesia
* Skin or scalp condition precluding use of external audio processor

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Functional gain | Up to six (6) months post-activation
  Postoperative improvement in aided soundfield thresholds compared to preoperative unaided soundfield thresholds
Adverse events | Up to six (6) months post-activation
  Number and proportion of subjects experiencing serious device- and surgery-related adverse events

SECONDARY OUTCOMES:
Word recognition score | Up to six (6) months post-activation
  Postoperative improvement on aided Consonant-Nucleus-Consonant (CNC) Words compared to preoperative unaided CNC word score
Unaided bone-conduction pure-tone average (BC-PTA) | Up to three (3) months post-activation
  Postoperative shift in unaided bone-conduction BC-PTA compared to preoperative unaided BC-PTA
Post-intervention quality-of-life questionnaire | Up to six (6) months post-activation
  Total and subscale scores on Glasgow Children's Benefit Inventory

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Colorado Health/Children's Hospital of Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - University Hospital Newark/Rutgers New Jersey Medical School, Newark, New Jersey
  - University of North Carolina, Chapel Hill, North Carolina
  - The Ohio State University/Nationwide Children's Hospital, Columbus, Ohio
  - University of Utah Health/Primary Children's Hospital, Salt Lake City, Utah